CLINICAL TRIAL: NCT06030141
Title: Investigation of the Effect of Nigella Sativa Oil and Sesame Oil in Preventing Phlebitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, BURCU NAL, LECTURER, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KSBUHSU
Record Dates: First submitted 2023-08-15; First posted 2023-09-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Phlebitis; Peripheral Venous Catheterization
Keywords: Phlebitis; nigella sativa oil; sesame oil; Peripheral Venous Catheterization
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Intervention Model Description: In this study, catheter application and follow-up will be carried out by the researcher Burcu Nal, and phlebitis evaluation will be made by a specialist nurse other than the researcher. Patients will be aware that they are included in the study, but they will be blinded as one of the oils applied in the care they will be given will be used by hiding the information of which group they are in. In order to prevent bias, patients will be included in the study groups according to the assignment made from the Randomizer.org program. Since the data will be transferred to the SPSS program and the analysis will be done by an independent statistician, the bias will also be controlled in the data evaluation process.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nigella sativa oil application group (Experimental): Peripheral venous catheter is applied under aseptic conditions. In order to easily see whether phlebitis occurs in the catheter area, the area where the catheter is inserted is covered with a Tegaderm transparent film cover and the catheter is fixed. Determine the distal peripheral venous catheter (3.2 cm length from the entry point for catheter 20) An area of 10 cm will be determined from the distal of the catheter. Nigella sativa oil is dripped 5 drops on a 10 cm area.
  The dripped oil is applied without massaging, Nigella Sativa oil will be applied to the patients in the application group before the start of amiodarone infusion and at 6-hour intervals. The patients in all groups will be evaluated with the GIFTS scale for phlebitis every hour for the first 25 hours from the time of opening the catheter, and every 6 hours for the next 48 hours.
  Interventions: Other: nigella sativa oil application
- Sesame oil application group (Experimental): Peripheral venous catheter is applied under aseptic conditions. In order to easily see whether phlebitis occurs in the catheter area, the area where the catheter is inserted is covered with a Tegaderm transparent film cover and the catheter is fixed. Determine the distal peripheral venous catheter (3.2 cm length from the entry point for catheter 20) An area of 10 cm will be determined from the distal of the catheter. Sesame oil is dripped 5 drops on a 10 cm area.
  The dripped oil is applied without massaging, The dripped oil is applied without massaging, Sesame oil will be applied to the patients in the application group before the start of amiodarone infusion and at 6-hour intervals. The patients in all groups will be evaluated with the GIFTS scale for phlebitis every hour for the first 25 hours from the time of opening the catheter, and every 6 hours for the next 48 hours.
  Interventions: Other: sesame oil application
- control group (No Intervention): Peripheral venous catheter is applied under aseptic conditions. In order to easily see whether phlebitis occurs in the catheter area, the area where the catheter is inserted is covered with a Tegaderm transparent film cover and the catheter is fixed. No oil application will be made. The patients in all groups will be evaluated with the GIFTS scale for phlebitis every hour for the first 25 hours from the time of opening the catheter, and every 6 hours for the next 48 hours.

INTERVENTIONS:
Other: sesame oil application — sesame oil application
  Arms: Sesame oil application group
Other: nigella sativa oil application — nigella sativa oil application
  Arms: nigella sativa oil application group

SUMMARY:
Phlebitis is an inflammatory reaction of the venous system and surrounding tissues that may be associated with mechanical, chemical or infectious microorganisms; It is the most common complication of intravenous injection. Symptoms of phlebitis; local pain, swelling, warmth, erythema, tenderness; prominent redness and palpable firmness and purulent discharge along the vascular access.

Phlebitis is the most important peripheral intravenous catheter-related complication and is seen in 0.1%- 63.3% of patients with peripheral intravenous catheters. Intravenous amiodarone is an important treatment for arrhythmias. However, peripheral infusion causes direct irritation of the vessel walls. Intravenous amiodarone is one of the most widely used antiarrhythmics for the treatment of atrial fibrillation with rapid ventricular response.

However, peripheral infusion of amiodarone usually causes pain during the infusion followed by phlebitis. Peripheral intravenous infusion of amiodarone associated with phlebitis is common in clinical practice, with an incidence of 5% to 65%.

Herbal treatment is a popular method in recent years In recent studies to prevent phlebitis, it has been determined that topical application of sesame oil and black cumin oil is effective in preventing phlebitis.

Sesame oil has antioxidant, anti-inflammatory and antibacterial properties and contains several lignans such as sesamin and sesaminol that inhibit inflammation, including interleukin 8 and endothelin 1. The therapeutic properties of black seed oil are due to the presence of phenolic compounds, especially thymoquinone. The anti-inflammatory mechanism of action of black seed oil occurs by inhibiting cyclo-oxygenase and 5-lipoxygenase pathways and preventing the production of thromboxane B2 and leukotriene B4.

There is no study in the literature comparing the effects of sesame oil and black cumin oil to prevent phlebitis.

DETAILED DESCRIPTION:
hlebitis is an inflammatory reaction of the venous system and surrounding tissues that may be associated with mechanical, chemical or infectious microorganisms; It is the most common complication of intravenous injection. Symptoms of phlebitis; local pain, swelling, warmth, erythema, tenderness; prominent redness and palpable firmness and purulent discharge along the vascular access.

Phlebitis is the most important peripheral intravenous catheter-related complication and is seen in 0.1%- 63.3% of patients with peripheral intravenous catheters. Intravenous amiodarone is an important treatment for arrhythmias. However, peripheral infusion causes direct irritation of the vessel walls. Intravenous amiodarone is one of the most widely used antiarrhythmics for the treatment of atrial fibrillation with rapid ventricular response.

However, peripheral infusion of amiodarone usually causes pain during the infusion followed by phlebitis. Peripheral intravenous infusion of amiodarone associated with phlebitis is common in clinical practice, with an incidence of 5% to 65%.

Herbal treatment is a popular method in recent years In recent studies to prevent phlebitis, it has been determined that topical application of sesame oil and black cumin oil is effective in preventing phlebitis.

Sesame oil has antioxidant, anti-inflammatory and antibacterial properties and contains several lignans such as sesamin and sesaminol that inhibit inflammation, including interleukin 8 and endothelin 1. The therapeutic properties of black seed oil are due to the presence of phenolic compounds, especially thymoquinone. The anti-inflammatory mechanism of action of black seed oil occurs by inhibiting cyclo-oxygenase and 5-lipoxygenase pathways and preventing the production of thromboxane B2 and leukotriene B4.

There is no study in the literature comparing the effects of sesame oil and black cumin oil to prevent phlebitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* IV amiodarone treatment was started,
* PIC applied to the cephalic or basilic vein,
* Number 20 catheter is preferred in PIC application,
* At least primary school graduate and can speak Turkish,
* Patients who voluntarily agree to participate in the study will be included in the study.

Exclusion Criteria:

* Diagnosed with active phlebitis,
* Having a diagnosis of mental illness or communication problems,
* Hearing and vision problems,
* Skin integrity is impaired,
* Having a body temperature above 38.5 Cº,
* Stating that he is allergic to sesame oil and black cumin oil,
* Receiving irritant medication or liquid other than Amiodarone through the catheter,
* Receiving long-term IV therapy from cephalic or basilic veins,
* Mastectomy surgery, fistula,
* who have been diagnosed with SVO,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
visual infusion phlebitis scale | Phlebitis formation is not expected during the follow-up period (72 hours) in the nigella sativa oil applied group.
  The scale has Turkish validity and durability.No change is expected in the Visual Infusion Phlebitis Scale score (2 points and above) in the sesame oil administration group (36 individual)
visual infusion phlebitis scale | Phlebitis formation is not expected during the follow-up period (72 hours) in the nigella sativa oil applied group.
  The scale has Turkish validity and durability.No change is expected in the Visual Infusion Phlebitis Scale score (2 points and above) in the nigella sativa oil administration group (36 individual)
visual infusion phlebitis scale | Phlebitis formation is expected during the follow-up period (72 hours) in the control group.
  The scale has Turkish validity and durability.Changes in the Visual Infusion Phlebitis Scale score (2 points and above) are expected in the control group (36 individuals).

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University Training and Research Hospital, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No